CLINICAL TRIAL: NCT03844347
Title: Well-being and Stress Control After Colorectal Surgery
Acronym: C-Bien
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7317
Record Dates: First submitted 2019-02-11; First posted 2019-02-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Patients with Colorectal Cancer; Surgery
Keywords: Colorectal cancer; Well-being; Stress; Recovery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C-Bien (Experimental)
  Interventions: Behavioral: Stress management sessions
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Stress management sessions — Stress management sessions are proposed to the patients and consist of small exercises focused on breathing and bodily sensations. Each accompanying person has access to different exercises. The sessions are adapted to the state of the patient to promote his well-being, before or after his/her operation. The duration of a preoperative session is 1 hour, the duration of the postoperative sessions is 15 minutes.
  Arms: C-Bien

SUMMARY:
The criteria usually considered to evaluate the quality of life are the presence or absence of a stomy, alteration of the transit or the sexual dysfunctions. Quality of life has been improved by introducing an Enhanced Postoperative Rehabilitation Program After Surgery (ERAS). It is a multidisciplinary medical and paramedical care aimed at minimizing the sources of stress allowing a significant reduction in postoperative complications and length of stay.

However, the emotional feelings of patients, their fatigue, the quality of their relationships with others and their experience of the disease are not usually considered. Nevertheless, these criteria influence the quality of life and constitute the fundamental bases of the psychological well-being, essential in the recovery processes.

We propose to enrich the ERAS program by introducing an individualized support of well-being and stress management aimed at increasing the quality of life of patients. The purpose is to make the patient more autonomous by allowing him/her, to implement stress management exercises.

The main goal of the project is to improve the psychological well-being of patients operated on for colorectal cancer by offering stress management sessions in order to promote postoperative rehabilitation.

The secondary objectives are to demonstrate the impact of stress management sessions on the length of stay and to study the link between the efficiency of these sessions and the quality of life of patients before the surgery.

ELIGIBILITY:
Inclusion criteria:

* Patient undergoing colorectal cancer surgery
* Regulated surgery
* With or without radiation treatment and / or preoperative chemotherapy.
* Patient benefiting from a social protection scheme

Exclusion criteria:

-- Limitation of linguistic or cognitive abilities interfering with the understanding of the study protocol

* Absence of the consent form of the study
* Emergency surgery
* Stomy closure
* Patient diagnosed psychotic.
* Patient with "psychiatric disorder" left to the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy Colorectal | 7 days before surgery
  The general well-being questionnaire (FACTC), validated with patients with colorectal cancer, which will allow us to measure the subjective feelings (physical, emotional and social well-being) of patients before hospitalization and on leaving the hospital
Functional Assessment of Cancer Therapy Colorectal | 5 days after surgery (the day of hospital leaving)
  The general well-being questionnaire (FACTC), validated with patients with colorectal cancer, which will allow us to measure the subjective feelings (physical, emotional and social well-being) of patients before hospitalization and on leaving the hospital
Manifestations of Psychological Well-being Measurement | 7 days before surgery
  Patient general quality of life measurement
Manifestations of Psychological Well-being Measurement | 5 days after surgery (the day of hospital leaving)
  Patient general quality of life measurement

SECONDARY OUTCOMES:
Fatigue measure | 7 days before surgery
  The MFI (Multidimensional Inventory of Fatigue)
Fatigue measure | 5 days after surgery (the day of hospital leaving)
  The MFI (Multidimensional Inventory of Fatigue)
Fatigue measure | 1 day after surgery up to 5 days after surgery (the day of hospital leaving)
  the BFI (Brief Fatigue Inventory) assess the physical and mental fatigue
Sleep quality assessment | 7 days before surgery
  Assessed with the Pittsburgh Sleep Quality Index score
Sleep quality assessment | 1 day after surgery up to 5 days after surgery (the day of hospital leaving)
  Assessed with the Pittsburgh Sleep Quality Index score
Pain assessment | 7 days before surgery
  Evaluation of the subjective pain sensation with the EVA score
Pain assessment | 1 day after surgery up to 5 days after surgery (the day of hospital leaving)
  Evaluation of the subjective pain sensation with the EVA score
Physical activity evaluation | 1 day after surgery up to 5 days after surgery (the day of hospital leaving)
  Actimetric evaluation: measurement of sleep phases and number of steps (Actiwatch AW7)

CONTACTS AND LOCATIONS:
Overall Officials: Benoît ROMAIN, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No